CLINICAL TRIAL: NCT01403103
Title: Evaluation of the Effect of 25-OH-Vitamin D3 Therapy on 15-Prostaglandin Dehydrogenase Expression in Primary Tumor and Normal Colorectal Mucosa in Patients With Colorectal Cancer
Brief Title: Cholecalciferol(25-[OH]-Vitamin D) in Treating Patients With Colorectal Cancer
Status: Withdrawn | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Slow Accrual
Sponsor: Case Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CASE2210; NCI-2011-01280 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2011-07-25; First posted 2011-07-27 (Estimated); Last update posted 2014-01-17 (Estimated); Status verified 2014-01

CONDITIONS: Mucinous Adenocarcinoma of the Colon; Mucinous Adenocarcinoma of the Rectum; Signet Ring Adenocarcinoma of the Colon; Signet Ring Adenocarcinoma of the Rectum; Stage I Colon Cancer; Stage I Rectal Cancer
MeSH Terms: conditions — Colonic Neoplasms; Rectal Neoplasms | interventions — Cholecalciferol; Biopsy; Enzyme-Linked Immunosorbent Assay; Reverse Transcriptase Polymerase Chain Reaction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (chemoprevention) (Experimental): Patients receive cholecalciferol orally (PO) 7 days prior to scheduled surgery or endorectal ultrasound. Patients with sigmoid colon cancer or clinical stage I rectal cancer would proceed with surgical resection without preceding chemoradiation and will have a portion of normal colorectal mucosa and tumor tissue obtained for research purposes.
  Interventions: Dietary Supplement: cholecalciferol; Procedure: biopsy; Genetic: protein expression analysis; Other: enzyme-linked immunosorbent assay; Other: laboratory biomarker analysis; Genetic: reverse transcriptase-polymerase chain reaction

INTERVENTIONS:
Dietary Supplement: cholecalciferol — Given PO
  Other Names: Calciol; Vitamin D3
Procedure: biopsy — Correlative studies
  Other Names: biopsies
Genetic: protein expression analysis — Correlative studies
Other: enzyme-linked immunosorbent assay — Correlative studies
  Other Names: ELISA
Other: laboratory biomarker analysis — Correlative studies
Genetic: reverse transcriptase-polymerase chain reaction — Correlative studies
  Other Names: RT-PCR

SUMMARY:
This pilot clinical trial studies cholecalciferol in treating patients with colorectal cancer. The use of cholecalciferol may slow disease progression in patients with colorectal cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To compare the expression of 15-hydroxyprostaglandin dehydrogenase (PGDH) messenger ribonucleic acid (mRNA) and protein levels in tumor tissue at baseline and after treatment with 25-hydroxy (OH)-vitamin D3 (cholecalciferol).

II. To compare the expression of 15-PGDH mRNA and protein levels in normal colorectal mucosa at baseline and following treatment with 25-OH-vitamin D3.

SECONDARY OBJECTIVES:

I. To compare the expression of cyclooxygenase (COX)-1 and COX-2 mRNA in tumor tissues at baseline and after treatment with 25-OH-vitamin D3.

II. To compare levels of prostaglandin E2 (PGE2) in tumor tissue at baseline and after treatment with 25-OH-vitamin D3.

III. To compare the expression of COX-1 and COX-2 mRNA in normal colorectal mucosa at baseline and after treatment with 25-OH-vitamin D3.

IV. To compare levels of PGE2 in normal colorectal mucosa at baseline and after treatment with 25-OH-vitamin D3.

V. To evaluate the tolerability of a single 100,000 international unit (IU) dose of 25-OH-vitamin D3.

OUTLINE:

Patients receive cholecalciferol orally (PO) 7 days prior to scheduled surgery or endorectal ultrasound. Patients are only followed through surgery or endorectal ultrasound. In case of a vitamin-D-related toxicity, the patient will be followed for resolution of the toxicity, up to 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a suspected diagnosis of adenocarcinoma of the rectum or sigmoid colon (e.g. based on appearance of mass or histology) referred to colorectal surgery who are expected to undergo routine proctosigmoidoscopy or flexible sigmoidoscopy in the surgeon's office as well as resection and/or endorectal ultrasound (EUS) as part of their routine care
* The tumor must be accessible for biopsy and suitable for multiple biopsies
* Eastern Cooperative Oncology Group (ECOG) performance status of =< 2
* Able to understand and willing to sign written informed consent document

Exclusion Criteria:

* Prior anti-cancer therapy for this cancer such as chemotherapy, biologic therapy, immune therapy or radiation therapy
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Unable to swallow capsules
* Underlying condition that will interfere with absorption of orally ingested vitamin D, e.g., untreated fat malabsorption
* History of allergic reaction to cholecalciferol or other vitamin D preparations
* EXCLUSION CRITERIA FOR DOSING VITAMIN D:
* Elevated ionized calcium
* Primary hyperparathyroidism
* Renal failure with estimated glomerular filtration rate < 20 mL/min/1.73m^2 as calculated using the Modification of Diet in Renal Disease (MDRD) study equation for the isotope dilution mass spectrometry (IDMS) - traceable creatinine methods reported by University Hospital Case Medical Center (UHCMC) laboratory (due to less active formation of 1,25 hydroxyvitamin D due to less hydroxylase)
* Serum 25-OH-vitamin D > 40 ng/ml

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-04; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Comparison of the expression of 15-PGDH mRNA and protein levels in tumor tissue | 7-14 days after treatment
  An increase in 15-PGDH expression will be defined as at least a 100% increase in mRNA by real-time reverse transcriptase (RT)-polymerase chain reaction (PCR) compared to baseline. Expression of 15-PGDH protein via ELISA in normal and tumor tissue at baseline and following treatment with vitamin D, as well as the absolute and fold changes will be summarized with descriptive statistics (e.g., mean, median, standard deviation, and interquartile range) and using box plots. In addition, 95% confidence intervals for the mean absolute and fold-changes in 15-PGDH levels will be calculated.
Comparison of the expression of 15-PGDH mRNA and protein levels in normal colorectal mucosa | 7-14 days after treatment
  An increase in 15-PGDH expression will be defined as at least a 100% increase in mRNA by real-time reverse transcriptase (RT)-polymerase chain reaction (PCR) compared to baseline. Expression of 15-PGDH protein via ELISA in normal and tumor tissue at baseline and following treatment with vitamin D, as well as the absolute and fold changes will be summarized with descriptive statistics (e.g., mean, median, standard deviation, and interquartile range) and using box plots. In addition, 95% confidence intervals for the mean absolute and fold-changes in 15-PGDH levels will be calculated.

SECONDARY OUTCOMES:
Comparison of the expression of COX-1 and COX-2 mRNA in tumor tissues | 7-14 days after treatment
Comparison of levels of PGE2 in tumor tissue | 7-14 days after treatment
Comparison of the expression of COX-1 and COX-2 mRNA in normal colorectal mucosa | 7-14 days after treatment
Comparison of levels of PGE2 in normal colorectal mucosa | 7-14 days after treatment
Number of patients with grade 3 related toxicities of a single 100,000 IU dose of 25-OH-vitamin D3 | 18-25 days after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Smitha Krishnamurthi, MD, Principal Investigator — Case Medical Center, University Hospitals Seidman Cancer Center, Case Comprehensive Cancer Center; Matthew Kalady, MD, Principal Investigator — Cleveland Clinic Taussig Cancer Institute, Case Comprehensive Cancer Center